CLINICAL TRIAL: NCT04650620
Title: Open, Non-comparative Study to Evaluate the Performance and Safety of the Medical Device Plenhyage® (Polymerized Polynucleotides Dermal Filler) in the Correction of Wrinkles and Improving the Skin Tones and Irregularities (Atrophies) of the Skin Surface in Neck, Abdomen, Thighs, and Buttocks
Brief Title: Study to Evaluate the Performance and Safety of the Medical Device Plenhyage®
Acronym: Plenhyage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.A. Istituto Ricerche Applicate S.p.A. (Network)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OPIRA/0419/MD
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Wrinkle

STUDY DESIGN:
Intervention Model Description: 20 patients will be administered Plenhyage® thin for the treatment of mild wrinkles;
  20 patients will be administered Plenhyage® medium for the treatment of moderate wrinkles;
  20 patients will be administered Plenhyage® strong for improving the skin tones and irregularities (atrophies) of the skin surface in neck, abdomen, thighs and buttocks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Plenhyage® thin (Experimental): Plenhyage® thin for the treatment of mild wrinkles;
  Interventions: Device: Plenhyage® thin
- Plenhyage® medium (Experimental): Plenhyage® medium for the treatment of moderate wrinkles;
  Interventions: Device: Plenhyage® medium
- Plenhyage® strong (Experimental): Plenhyage® strong for improving the skin tones and irregularities (atrophies) of the skin surface in neck, abdomen, thighs and buttocks
  Interventions: Device: Plenhyage® strong

INTERVENTIONS:
Device: Plenhyage® thin — 0.75%
  Arms: Plenhyage® thin
Device: Plenhyage® medium — 2%
  Arms: Plenhyage® medium
Device: Plenhyage® strong — 2.5%
  Arms: Plenhyage® strong

SUMMARY:
The Research Question of the present study is the following: in a population of men and women affected by face wrinkles and skin tones and irregularities (atrophies) of the skin surface in neck, abdomen, thighs and buttocks, will Plenhyage® significantly decrease the appearance of treated areas, results observed after 8 and 12 weeks?

DETAILED DESCRIPTION:
Open, non-comparative, interventional, multicenter study with the total number of screened subjects of 66 (60 evaluable subjects +6 potential screening failure):

* 20 patients will be administered Plenhyage® thin for the treatment of mild wrinkles;
* 20 patients will be administered Plenhyage® medium for the treatment of moderate wrinkles;
* 20 patients will be administered Plenhyage® strong for improving the skin tones and irregularities (atrophies) of the skin surface in neck, abdomen, thighs and buttocks;

ELIGIBILITY:
Inclusion Criteria:

1. Men or women with age ≥ 30 and ≤ 67 years;
2. Subjects presenting a score of 2 (mild facial wrinkles) for Plenhyage® thin, 3 (moderate facial wrinkles) for Plenhyage® medium on the Wrinkles Severity Ranking Scale (WSRS) seeking skin imperfections treatment;
3. Subjects presenting a ANA score < 5 seeking treatment for defect and irregularities (atrophies) of the skin surface in neck, abdomen, thighs or buttocks for Plenhyage® strong;
4. Subjects who agree to discontinue all dermatological treatment and procedures during the study.
5. Subjects willing to provide signed informed consent to clinical investigation participation.
6. Able to communicate adequately with the Investigator and to comply with the requirements for the entire study.

Exclusion Criteria:

1. Use of aspirin and antiplatelet agents a week prior to treatment;
2. Subjects with history of allergy or hypersensitivity to polymerized polynucleotides or to other ingredients of the dermal filler or hypersensitivity skin reaction to the investigational device based on intradermal test results at visit 1.
3. Subjects with any dermal systemic pathologies, such as systemic lupus erythematosus, psoriasis, scleroderma etc.;
4. Subjects presenting bleeding disorders in the past or present;
5. Subjects taking or having indications for anticoagulant therapy;
6. Use of concomitant treatments or procedures aimed to improve skin rejuvenation over the last six months before the clinical investigation enrolment, such as chemical peeling, dermabrasion, laser resurfacing;
7. Subjects suffering from infectious diseases including herpes simplex virus infection, active hepatitis or human immunodeficiency virus;
8. Subjects suffering from eczema, acne and keloids;
9. Subjects with any cutaneous manifested infection, disease or alteration;
10. Subjects at risk in term of precautions, warnings and contra-indications referred in the package insert of the clinical investigation device;
11. Subjects with any facial aesthetic surgery in the preceding 12 months before the clinical investigation enrolment;
12. Subjects with any active irritation or inflammation in the target areas of injection;
13. Subjects who received botulinum toxin A injections in the face in the preceding 6 months;
14. Subjects unlikely to cooperate in the clinical investigation or to comply with the treatment or with the clinical investigation visits;
15. Pregnant woman, lactating woman, and man or woman of childbearing potential who is planning a pregnancy or is unwilling to use appropriate methods of contraception* during the study, *Methods of contraception: hormonal contraceptive, intrauterine device or intrauterine system, double barrier method (condom with spermicide/diaphragm or cervical cap with spermicide), surgical sterilization (vasectomy, tubal ligation, etc.).
16. Subjects with illness, or other medical condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the study.
17. Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days.

Ages: 30 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Wrinkle Severity Rating Scale score evaaluated by the Investigator | 12 weeks
  The WSRS score performed by Investigator have been chosen as a primary efficacy outcome to measure the performance of the Plenhyage® thin and medium. The scale has 5 grades: 1 absent, 2 mild, 3 moderate, 4 severe, 5 extreme, where 1 absent represents no visible folds and 5 extreme represent extreme deep and long folds.
Aesthetic Numeric Scale evaluated by the Investigator | 12 weeks
  The ANA score will be evaluated on a point scale from 0 to 10 where:
  0 - Insufficient
  1. - Unsatisfied
  2. - Poor
  3. - Sufficient
  4. - Neutral
  5. - Agreed
  6. - Satisfied
  7. - As requested
  8. - Perfect
  9. - Harmonic
  10. - Highly satisfied The best score for ANA score is 10 highly satisfied and the worst outcome is 0 insufficient

SECONDARY OUTCOMES:
WSRS score evaluated by the subject | 12 weeks
  The WSRS score performed by subject has been chosen as a secondary efficacy outcome to measure the performance of the Plenhyage® thin and medium. The scale has 5 grades: 1 absent, 2 mild, 3 moderate, 4 severe, 5 extreme, where 1 absent represents no visible folds and 5 extreme represent extreme deep and long folds.
Global Aesthetic Improvement Scale | 12 weeks
  Subjects will evaluate their skin appearance change compared to before the treatment, as follows:
  Very Much Improved (1) = Optimal cosmetic result; Much Improved (2) = Market improvement in appearance but not completely optimal. A touch-up would slightly improve the result; Improved (3) = Obvious improvement in appearance from the initial condition, but a touch-up or re-treatment is indicated; No Change (4) = The appearance is essentially the same as the original condition; Worse (5) = The appearance is worse than the original condition.
Treatment satisfaction | 12 weeks
  Treatment satisfaction will be assessed by the subject at 4, 8 and 12 weeks using a 4-point scale: very satisfied, satisfied, moderate and not satisfied;
Investigator Global Assessment of Performance | 12 weeks
  Investigator Global Assessment of Performance (IGAP) Investigator will make photographs at every visit (1, 2, 3, 4 and 5) of the area treated in order to evaluate the performance of the treatment at visit 5 using a 4-point scale: 1= very good performance, 2 = good performance, 3 = moderate performance and 4 = poor performance;
Investigator Global Assessment of Safety | 12 weeks
  Investigator Global Assessment of Safety (IGAS) will be reported using the 4-point scale: 1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety. IGAS will be evaluated by the Investigator at Final visit (12 weeks), only;
Patient Global Assessment of Safety | 12 weeks
  Patient Global Assessment of Safety (PGAS) will be reported by the subject at the last visit using the 4-point scale: 1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety. PGAS will be evaluated by the patient at Final visit (12 weeks), only.

CONTACTS AND LOCATIONS:
Locations (1):
- SCM Dr. Rosu, Timișoara, Timiș County, Romania